CLINICAL TRIAL: NCT05307640
Title: Caregiver Wellness After Traumatic Brain Injury (CG-WELL): An Intervention Designed to Promote Well-being in Caregivers of Acute Moderate to Severe Traumatic Brain Injuries
Acronym: CG-Well
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natalie Kreitzer (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Natalie Kreitzer, Associate Professor Emergency Medicine, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-1198
Record Dates: First submitted 2022-03-14; First posted 2022-04-01 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Trauma, Brain
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CG-Well (Experimental): CG-Well is a web & phone based psychosocial intervention that teaches caregivers how to obtain information, education & support
  Interventions: Behavioral: CG-Well
- Information Support and Referral (Placebo Comparator): Attention control group that receives phone calls and modules from the Brain Injury Association of America.
  Interventions: Behavioral: Information Support & Referral (ISR)

INTERVENTIONS:
Behavioral: CG-Well — CG-Well is a web & phone based psychosocial intervention that teaches caregivers how to obtain information, education & support
  Arms: CG-Well
Behavioral: Information Support & Referral (ISR) — Attention control group that receives phone calls and modules from the Brain Injury Association of America.
  Arms: Information Support and Referral

SUMMARY:
After injury, survivors of msTBI depend on informal family caregivers. Upwards of 77% of family caregivers experience poor outcomes, such as adverse life changes, poor health related quality of life, and increased depressive symptoms. Caregivers frequently report minimal support or training to prepare them for their new role. Periods of care transitions, such as ICU discharge, are most difficult. The majority (93%) of previously developed caregiver and caregiver/survivor dyad interventions after msTBI focus on providing information or practical skills to either survivors, or to long-term caregivers (>6 months post injury), rather than education, support, and skill-building that the new caregiver may use proactively that will benefit the dyad acutely after injury. The Aims of this proposal are to: (1) Determine feasibility, satisfaction, and data trends of CG-Well; and (2) Understand how baseline psychosocial risk factors affect response to CG-Well compared to an Information, Support, and Referral control group. To accomplish this, I will first enroll 6-10 caregivers and tailor CG-well until each finds the intervention acceptable, appropriate, and feasible. I will then enroll 100 (50/group) dyads and determine satisfaction ratings, recruitment, retention, and treatment fidelity of CG-Well. Additionally, I will determine if caregivers report reductions in depressive symptoms and improvements in life changes as a result of improvements in task difficulty and threat appraisal in CG-Well compared to ISR at six months. Information obtained in Aims 1 and 2 will be used to plan a larger Phase III trial of CG-Well. Completing these Aims and the training plan will improve outcomes of caregivers and downstream outcomes of survivors of msTBI, and provide me with the skillset necessary to become an independent researcher who can develop and test high-impact, high-fidelity, sustainable interventions.

ELIGIBILITY:
Inclusion criteria:

* Survivor and caregiver ≥18 years old
* Survivor GCS 3-12 after resuscitation
* Survivor < 2 weeks post injury
* English Speaking - survivor and caregiver

Exclusion criteria:

* Patient not expected to survive.
* Pregnant - survivor or caregiver
* Prisoner - survivor or caregiver
* History of pre-existing condition that would interfere with follow-up in caregiver or survivor (e.g., substance abuse, alcoholism, end-stage cancers)
* Major prior debilitating neurological or mental health disorder in caregiver or survivor (e.g., schizophrenia, bipolar, stroke, dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Intervention Satisfaction | 6 months
  Scale Title: Caregiver Intervention Satisfaction Scale. Likert's scale of usability, ease of use, and acceptability of INR or CG-Well A higher score indicates greater satisfaction; 1-5 scale (strongly disagree=1; strongly agree=5)

SECONDARY OUTCOMES:
Brief Symptom Inventory-18 (BSI-18) | 6 months
  Quantifies symptoms of somatization, depression, and anxiety. The BSI-18 consists of 18 items on a 5-point (0-4) Likert scale and is designed to assess current psychological distress (over the past 7 days). In addition to a total score, referred to as the Global Severity Index (GSI; max = 72), a separate score can be calculated on a depressive subscale: with six questions contributing to the subscale (max = 24). Raw scores will be converted to t-scores. Higher scores reflect greater distress.
Bakas Caregiver Outcomes Scale (BCOS) | 6 months
  Measures life changes specifically resulting from providing care, such as negative social, emotional, health-related, financial wellbeing, level of energy, and role functioning effects. Each change is rated on a seven-point Likert scale (-3=changed for the worst to +3=changed for the best).
Oberst Caregiving Burden Scale | 6 months
  Measures time and difficulty associated with caregiving tasks, such as providing personal care, managing emotions of the TBI survivor, and dealing with finances. Task difficulty is measured on a seven-point Likert scale (-3 extremely difficult to +3 extremely easy), and time is rated on a five-point Likert scale (5 = great amount, 1 = none).
Appraisal of Caregiving Scale Threat Subscale | 6 months
  Measures the caregiver appraisal of their current situation (threat and worry) by focusing on perceived threat. The ACS uses a five-point Likert scale to determine stress in the current situation (5 = strongly agree, 1 = strongly disagree).
Feasibility of CG-Well (Recruitment) | up to 30 months
  Measurements of recruitment: Will look at how many caregivers were approached vs. consented.
Feasibility of CG-Well (Retention) | 6 months
  Measurements of Retention: Will look at how many caregivers were still active in the study at the 6 month mark.
Feasibility of CG-Well (Treatment Fidelity) | up to 36 months
  Measurements of Treatment Fidelity: We will report the proportion of participants who have all elements of fidelity checklist (Borrelli Treatment Fidelity Checklist: Checklist makes sure the following is completed: Standardized research coordinator training, Documentation of study activity at each session, Audio recorded calls, PI, mentor and third party coordinator review 20% of recorded sessions and Team meetings to discuss treats to fidelity.
  These checklists are reviewed on a weekly basis.
Feasibility of CG-Well (Number of Log Ins to the website) | up to 36 months
  Participant reported number of times they log into the study website each month.
  Reported during study visit calls.
Feasibility of CG-Well (Time that the participant spent in modules) | up to 36 months
  Participant reported length of time spent each month on the website or in modules.
  Reported during study visit calls.
Feasibility of CG-Well (Time spent in monthly phone calls with the study team) | up to 36 months
  Study phone calls are recorded and time stamped.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Kreitzer N, Fink S, Adeoye O, Kurowski G B, Wade S, Sucharew H, Bakas T. Caregiver Wellness after Traumatic Brain Injury (CG-Well): Protocol for a randomized clinical trial. Contemp Clin Trials Commun. 2024 Aug 24;41:101356. doi: 10.1016/j.conctc.2024.101356. eCollection 2024 Oct. PMID 39280784